CLINICAL TRIAL: NCT05504460
Title: A Randomized, Controlled Clinical Trial to Evaluate the Effectiveness and Safety of Hydrogen-Oxygen Generator With Nebulizer for Rehabilitation Treatment of Dysfunctions in Discharged Patients Who Are Previously Hospitalized Due to COVID-19
Brief Title: Hydrogen-Oxygen Generator With Nebulizer for Rehabilitation Treatment of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMS-H-03-104
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; AMS-H-03; Hydrogen-oxygen Gas
Keywords: COVID-19; Hydrogen-Oxygen Generator with Nebulizer; AMS-H-03; Hydrogen-oxygen Gas
MeSH Terms: conditions — COVID-19 | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: The test group will use the investigational device Hydrogen-Oxygen Generator with Nebulizer (manufactured by Shanghai Asclepius Meditec Co., Ltd.) + basic treatment (supportive treatment determined by the investigator based on the condition of the patients), and the control group will use basic treatment only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): The test group will use the investigational device Hydrogen-Oxygen Generator with Nebulizer (manufactured by Shanghai Asclepius Meditec Co., Ltd.) + basic treatment (supportive treatment determined by the investigator based on the condition of the patients)
  Interventions: Device: Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03; Other: basic treatment
- Control Group (Active Comparator): the control group will use basic treatment only
  Interventions: Other: basic treatment

INTERVENTIONS:
Device: Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03 — Treatments in the test group will lasts for 12 months, and symptomatic treatment will be provided based on the actual symptoms of the subjects. Subjects in the test group will be required to receive inhalation for at least 4 days every 7 days with at least 3780L inhaled every 7 days (It is recommended to inhale at least 540L per day; If the flow rate is 3L/min, it is recommended that the cumulative inhalation time should be at least 3 hours per day. If the flow rate is 1.5L/min, it is recommended that the cumulative inhalation time should be at least 6 hours per day).
  Arms: test group
Other: basic treatment — supportive treatment determined by the investigator based on the condition of the patients

SUMMARY:
This is a prospective, multicenter, randomized, controlled, superiority clinical trial, with the test group expected to be superior to the control group in the primary evaluation endpoints (changes in Borg score and PSQI index at 3 months after the start of the treatment). The test group will use the investigational device Hydrogen-Oxygen Generator with Nebulizer (manufactured by Shanghai Asclepius Meditec Co., Ltd.) + basic treatment (supportive treatment determined by the investigator based on the condition of the patients), and the control group will use basic treatment only, to evaluate of effectiveness and safety of the investigational device Hydrogen-Oxygen Generator with Nebulizer for rehabilitation treatment of dysfunctions in discharged patients who are previously hospitalized due to 2019 novel coronavirus pneumonia (COVID-19).

DETAILED DESCRIPTION:
A total of 216 eligible subjects will be randomly assigned to the test group and the control group in a 1:1 ratio to receive corresponding treatment (treatment in both groups will last for 12 months), and the subjects will then be followed up for 12 months from the start of treatment after enrollment.

All subjects enrolled in this study will receive seven visits, including the screening visit (within 14 days before the enrollment), randomization and treatment visit (Day 0), visits at 1 month after the start of the treatment (± 7 days), 2 months after the start of the treatment (± 7 days), 3 months (± 14 days) after the start of the treatment, 6 months (± 14 days) after the start of the treatment, and 12 months (± 30 days) after the start of the treatment.

The following indicators of the two groups will be collected and analyzed in this study: the primary effectiveness evaluation indicator: changes in Borg score and PSQI index at 3 months after the start of the treatment; secondary effectiveness evaluation indicators: 1) Pulmonary function assessment indicators (forced expiratory volume in one second [FEV1], ratio of forced expiratory volume in one second to forced vital capacity [FEV1/FVC], 25/50/75% maximal mid expiratory flow [MMEF 25/50/75], and fractional exhaled nitric oxide [FeNO]); 2) Lung imaging changes; 3) Neurological and psychological function assessment indicators (Mini-Mental State Examination Scale [MMSE] score, Generalized Anxiety Disorder Scale [GAD-7] score, Depression Screening Scale [PHQ-9] score, Post-Traumatic Stress Disorder Checklist [PCL-C]); 4) Inflammatory indicators (neutrophil-to-lymphocyte ratio [NLR], C-reactive protein [CRP], interleukin-6 [IL-6]); 5) Evaluation of device usability, and the safety evaluation indicators: incidence of AEs and SAEs, and incidence of device deficiencies.

When all enrolled subjects have completed the follow up at 3 months after the start of the treatment, an analysis will be performed for application to the National Medical Products Administration (NMPA) for registration of the investigational medical device, while the 6- and 12-month follow up will be continued spontaneously.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 and 75 years old (inclusive);
* Subjects previously hospitalized due to COVID-19, who are recovered and discharged with negative results for COVID-19 and released from quarantine;
* Known symptoms of respiratory dysfunctions (such as dyspnea), and / or neurological/psychological dysfunction (such as sleep disorders, anxiety, and depression) and / or somatic dysfunction (such as fatigue);
* Borg dyspnea or fatigue score before study treatment ≥ 1 (please refer to Appendix 2: Borg Scale for specific information), and PSQI score ≥ 2 (please refer to Appendix 3: PSQI Scale for specific information);
* Subjects who are willing to participate and provided written informed consent form.

Exclusion Criteria:

* Subjects with known malignant tumor;
* Subjects with known moderate or severe pulmonary infection;
* Subjects with mucosa injury in upper respiratory tract, for whom no inhalation treatment can be provided;
* Subjects who are intolerable to inhalation treatment;
* Subjects with moderate or severe disabilities;
* Subjects with mental disorders or cognitive impairment who are unable to provide consent;
* Subjects with neurological disease accompanied with sleep disorders for which medical intervention is provided before the diagnosis of COVID-19.
* Subjects with any immunodeficiency (for example, subjects requiring chronic treatment with any corticosteroid or other immunosuppressants) judged by the investigator;
* Allergy to any component of the investigational product that have contact with human body;
* Complicate severe cardiac, hepatic or renal insufficiency;
* Expected life expectancy < 1 year;
* Subjects who are participating in any other clinical study of any investigational drug or medical device;
* Pregnant or lactating women, or women who plan to become pregnant within the following one year;
* Any other condition judged as inappropriate to participate in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Borg score index from baseline at 3 months after the start of the study treatment. | Changes in Borg score assessed after the 6-minute walk test at 3 months (±7 days)
  after the start of the treatment compared to Borg score assessed after the 6-minute walk test before treatment in the test or the control group.
Changes in PSQI index from baseline at 3 months after the start of the study treatment. | Changes in PSQI index at 3 months (±7 days) after the start of the treatment of the subjects in the test group or the control group compared with that before treatment.
  Changes in PSQI index at 3 months (±7 days) after the start of the treatment of the subjects in the test group or the control group compared with that before treatment.

SECONDARY OUTCOMES:
Pulmonary function evaluation: FEV1 | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Pulmonary function evaluation: FEV1
Change in imaging evaluation | 3 months (±14 days), 6 months (±14 days, as needed), and 12 months (±30 days)
  It is defined as the change in lung imaging results evaluated by CT examination
Neurological and psychological function indicators including MMSE score | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Neurological and psychological function indicators including MMSE score
Inflammatory indicators, including NLR | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Inflammatory indicators, including NLR
Usability evaluation of the medical device | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  It is defined as the results of the evaluation on usability of the investigational medical device conducted according to the following table
Pulmonary function evaluation: FEV1/FVC | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Pulmonary function evaluation: FEV1/FVC
Pulmonary function evaluation: MMEF 25 | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Pulmonary function evaluation: MMEF 25
Pulmonary function evaluation: MMEF50 | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Pulmonary function evaluation: MMEF 50
Pulmonary function evaluation: MMEF 75 | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Pulmonary function evaluation: MMEF 75
Pulmonary function evaluation: FeNO | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Pulmonary function evaluation: FeNO
Neurological and psychological function indicators including GAD-7 score | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Neurological and psychological function indicators including GAD-7 score
Neurological and psychological function indicators including PHQ-9 score | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Neurological and psychological function indicators including PHQ-9 score
Neurological and psychological function indicators including PCL-C score | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Neurological and psychological function indicators including PCL-C score
Inflammatory indicators, including CRP | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Inflammatory indicators, including CRP
Inflammatory indicators, including IL-6 | 1 month (±7 days), 2 months (±7 days), 3 months (±14 days), 6 months (±14 days) and 12 months (±30 days)
  Inflammatory indicators, including IL-6

OTHER OUTCOMES:
AE/SAE percentage | through study completion, an average of 1 year
  AE/SAE percentage
Rate of device deficiency | through study completion, an average of 1 year
  Device deficiency refers to the unreasonable risks that may endanger human health and life safety in the normal use of the medical device during the clinical trial, such as label errors, quality problems and malfunctions.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sanyaolu A, Marinkovic A, Prakash S, Zhao A, Balendra V, Haider N, Jain I, Simic T, Okorie C. Post-acute Sequelae in COVID-19 Survivors: an Overview. SN Compr Clin Med. 2022;4(1):91. doi: 10.1007/s42399-022-01172-7. Epub 2022 Apr 6. PMID 35411333
- [Background] Huang L, Yao Q, Gu X, Wang Q, Ren L, Wang Y, Hu P, Guo L, Liu M, Xu J, Zhang X, Qu Y, Fan Y, Li X, Li C, Yu T, Xia J, Wei M, Chen L, Li Y, Xiao F, Liu D, Wang J, Wang X, Cao B. 1-year outcomes in hospital survivors with COVID-19: a longitudinal cohort study. Lancet. 2021 Aug 28;398(10302):747-758. doi: 10.1016/S0140-6736(21)01755-4. PMID 34454673
- [Background] Blomberg B, Mohn KG, Brokstad KA, Zhou F, Linchausen DW, Hansen BA, Lartey S, Onyango TB, Kuwelker K, Saevik M, Bartsch H, Tondel C, Kittang BR; Bergen COVID-19 Research Group; Cox RJ, Langeland N. Long COVID in a prospective cohort of home-isolated patients. Nat Med. 2021 Sep;27(9):1607-1613. doi: 10.1038/s41591-021-01433-3. Epub 2021 Jun 23. PMID 34163090
- [Background] Lopez-Leon S, Wegman-Ostrosky T, Perelman C, Sepulveda R, Rebolledo PA, Cuapio A, Villapol S. More than 50 long-term effects of COVID-19: a systematic review and meta-analysis. Sci Rep. 2021 Aug 9;11(1):16144. doi: 10.1038/s41598-021-95565-8. PMID 34373540
- [Background] Jennings G, Monaghan A, Xue F, Mockler D, Romero-Ortuno R. A Systematic Review of Persistent Symptoms and Residual Abnormal Functioning following Acute COVID-19: Ongoing Symptomatic Phase vs. Post-COVID-19 Syndrome. J Clin Med. 2021 Dec 16;10(24):5913. doi: 10.3390/jcm10245913. PMID 34945213
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Zheng ZG, Sun WZ, Hu JY, Jie ZJ, Xu JF, Cao J, Song YL, Wang CH, Wang J, Zhao H, Guo ZL, Zhong NS. Hydrogen/oxygen therapy for the treatment of an acute exacerbation of chronic obstructive pulmonary disease: results of a multicenter, randomized, double-blind, parallel-group controlled trial. Respir Res. 2021 May 13;22(1):149. doi: 10.1186/s12931-021-01740-w. PMID 33985501
- [Background] Guan WJ, Wei CH, Chen AL, Sun XC, Guo GY, Zou X, Shi JD, Lai PZ, Zheng ZG, Zhong NS. Hydrogen/oxygen mixed gas inhalation improves disease severity and dyspnea in patients with Coronavirus disease 2019 in a recent multicenter, open-label clinical trial. J Thorac Dis. 2020 Jun;12(6):3448-3452. doi: 10.21037/jtd-2020-057. No abstract available. PMID 32642277
- [Background] Liu ST, Zhan C, Ma YJ, Guo CY, Chen W, Fang XM, Fang L. Effect of qigong exercise and acupressure rehabilitation program on pulmonary function and respiratory symptoms in patients hospitalized with severe COVID-19: a randomized controlled trial. Integr Med Res. 2021;10(Suppl):100796. doi: 10.1016/j.imr.2021.100796. Epub 2021 Oct 29. PMID 34733607
- [Background] Xiao CX, Lin YJ, Lin RQ, Liu AN, Zhong GQ, Lan CF. Effects of progressive muscle relaxation training on negative emotions and sleep quality in COVID-19 patients: A clinical observational study. Medicine (Baltimore). 2020 Nov 20;99(47):e23185. doi: 10.1097/MD.0000000000023185. PMID 33217826